CLINICAL TRIAL: NCT01348880
Title: A Double-Blind Study to Evaluate the Pharmacodynamic Interaction Between 10 mg Vardenafil ODT (Orally Disintegrating Tablet) and Procardia XL® (Nifedipine GITS) in Elderly Male Patients With Both Hypertension and Erectile Dysfunction
Brief Title: Vardenafil ODT (Orally Disintegrating Tablet) - Nifedipine Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 15345
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Erectile Dysfunction
Keywords: drug-drug interaction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1 (Experimental)
  Interventions: Drug: Vardenafil ODT, (Staxyn, BAY38-9456)
- Arm2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil ODT, (Staxyn, BAY38-9456) — Single dose of 10 mg of vardenafil ODT, taken without water
  Arms: Arm1
Drug: Placebo — Single dose of placebo to match 10 mg vardenafil ODT. taken without water
  Arms: Arm2

SUMMARY:
The study will be conducted as a multi-center, randomized, double-blinded, placebo controlled, crossover design. The investigational drug (vardenafil ODT (Orally Disintegrating Tablet)/placebo) will be given as a single administration at a dose of 10 mg vardenafil ODT during Period 1 or 2; the blinded matching placebo will be given as a single administration during the opposing period. The random code will determine the order of active drug (vardenafil ODT) and placebo for each subject. Blood pressure and heart rate profiles will be recorded by automated device pre-dose for 8 hours post-dose during Periods 1 and 2. The non investigational drug product (vasodilator), Procardia XL, will be background treatment for hypertension, taken daily by each subject. All subjects must be stable on the vasodilator for at least 4 weeks prior to Day 1 of Period 1. Special conditions for this study include the requirement that all subjects will be male, are between the ages of 65 and 80 years, and will have a diagnosis of erectile dysfunction (ED), as well as hypertension. Planned sample size will be 40 subjects evaluable for the primary analysis. Of the 40 subjects valid for this analysis, 20 will be between the ages of 65 and 69 years, and 20 subjects will be between the ages of 70 and 80 years. The total duration of the study will be approximately one year from first subject treated to last subject treated, including replacement of any subjects who fail to complete both periods of crossover dosing.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria before being included in the treatment period i.e., before receiving any dose of the study related medication (Sponsor supplied Procardia XL, or vardenafil Orally Disintegrating Tablet (ODT) /placebo tablets):

* The informed consent must be signed before any study specific tests or procedures are done
* Male gender
* Diagnosis of both essential hypertension (HTN) and erectile dysfunction (ED)
* High blood pressure, or hypertension, is defined in an adult as a systolic pressure of 140 mm Hg or higher and/or a diastolic pressure of 90 mm Hg or higher. As stated in the current American Heart Association guidelines.
* Documented ED for more than 6 months according to the National Institutes of Health (NIH) Consensus statement (the inability to achieve or maintain penile erection sufficient for satisfactory sexual performance). The diagnosis for ED will be confirmed using the five-item version (Rosen RC) of the International Index of Erectile Function (IIEF-5), see Appendix 14.4. The total IIEF-5 score must be at least 8, and not exceed 19. Subjects must have used at least one Phosphodiesterase-5 (PDE-5) inhibitor, such as Viagra, Levitra or Cialis at some time prior to entry in this study.
* Age: 65 to 80 years (inclusive) at the first screening examination / visit
* Body mass index (BMI): above/equal 18 and below/equal 32 kg / m²

Exclusion Criteria:

Subjects are to be excluded from the study if they display any of the following criteria:

Medical and surgical history

* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal. This includes severe renal impairment (on dialysis or not) and moderate or severe hepatic disease.
* Known hypersensitivity to calcium channel blockers (active substances or excipients of the tablet preparations)
* Known hypersensitivity to PDE-5 inhibitors, such as Viagra, Levitra or Cialis (active substances or in some instances, excipients of the tablet preparations should be considered as possible allergens, e.g., lactose, aspartame)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Recent history (within 6 months) of myocardial infarction (MI), coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA), stenting, or cerebrovascular accident (CVA)
* Known left ventricular outflow syndrome (LVO)
* History of significant coronary artery disease, e.g., angina
* Congenital or acquired prolonged QT syndrome
* Congestive heart failure (CHF) [NYHA Class 3 or 4]
* History of adult epilepsy or other seizure disorders
* History of retinitis pigmentosa
* Use of any anti-hypertensive medication other than the calcium channel blocker, Procardia XL (nifedipine), supplied by the sponsor, during the study
* Any drug known to induce cytochrome P450 (CYP) enzymes (eg rifampicin, carbamazepine, phenytoin, bosentan, dexamethasone, barbiturates, St. John's Wort [hypericum perforatum])
* Any drug known to inhibit CYP enzymes: specifically potent or moderate cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors such as HIV protease inhibitors (e.g. ritonavir, indinavir, saquinavir, atazanavir), ketoconazole, itraconazole, clarithromycin and erythromycin
* Use of nitroglycerin or any form of nitrates is not allowed
* All alpha-blockers (e.g., Hytrin, Flomax, Uroxatral) are prohibited Electrocardiogram (ECG), blood pressure, heart rate
* Clinically relevant findings in the ECG such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTc-interval over 450 msec
* Systolic blood pressure below 110 or above 150 mmHg on anti-hypertensive therapy
* Diastolic blood pressure below 60 or above 95 mmHg on anti-hypertensive therapy
* Heart rate below 40 or above 95 beats / min on anti-hypertensive therapy
* Serum creatinine > 2.5 mg/dL at Screening
* HbA1c > 8% indicative of uncontrolled DM at Screening

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary pharmacodynamic variable (endpoint) is the placebo-corrected mean maximal decrease in supine systolic blood pressure from baseline (1 hour before dose) to within 8 hours of dosing with 10 mg ODT formulation of vardenafil HCl and nifedipine. | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine.

SECONDARY OUTCOMES:
Mean maximal decrease in standing SBP | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Mean maximal decrease in standing diastolic blood pressure (DBP) | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Mean maximal decrease in supine DBP | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Mean maximal orthostatic change in SBP (the supine SBP minus the standing SBP) | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Mean maximal increase in supine and standing heart rate | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Mean area under effect curve (AUEC) in standing and supine systolic and diastolic blood pressure, and heart rate | Up to 8 hours of combination dosing of vardenafil ODT and nifedipine
Safety parameters | up to end of study
  Safety parameters included physical examinations, adverse events, laboratory values, electrocardiogram, concomitant medications, and vital signs
Pharmacokinetics parameter | 1 and 2 weeks prior to the Day 1 dosing of the combination of nifedipine/vardenafil as well as at Visit 4 and Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Miami, Florida
  - Knoxville, Tennessee